CLINICAL TRIAL: NCT03071497
Title: Non-invasive Diagnostics of Iron Deficiency in Surgical Patients by Measuring Zinc Protoporphyrin-IX
Status: Completed | Type: Observational
Sponsor: Johann Wolfgang Goethe University Hospital (Other)
Collaborators: Ludwig-Maximilians - University of Munich (Other)
Responsible Party: Principal Investigator, Dr. Patrick Meybohm, M.D., Prof. Dr. Patrick Meybohm, Johann Wolfgang Goethe University Hospital
Other Study IDs: 468/16
Record Dates: First submitted 2017-02-25; First posted 2017-03-07 (Actual); Last update posted 2018-07-17 (Actual); Status verified 2018-07

CONDITIONS: Iron-deficiency; Anemia; Iron Deficiency Anemia
Keywords: Iron-deficiency; Anemia; Iron-deficiency Anemia; Zinc protoporphyrin
MeSH Terms: conditions — Anemia, Iron-Deficiency; Anemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study Group: Detecting iron deficiency using various methods. All patients that fit the inclusion criteria and are willing to participate in the study will be included in this group.
  Interventions: Diagnostic Test: Non-invasive analysis of Zinc protoporphyrin

INTERVENTIONS:
Diagnostic Test: Non-invasive analysis of Zinc protoporphyrin — In patients fitting the inclusion criteria Zinc protoporphyrin will be measured non-invasively as proxy for iron deficiency. Results will be compared to ZnPP reference values measured via HPLC and with spectroscopical measurements performed on whole blood as well as with blood values (HB, MCH, MCV, ferritin, CRP, transferrin saturation, soluble transferrin receptor) assessed during clinical routine.

SUMMARY:
* In approx. 40% of the incidences anemia is caused by iron deficiency (= ID). In turn, preoperative iron-deficiency anemia (= IDA) is associated with an increase in morbidity and mortality as well as with the need for a blood transfusion.
* A successful preoperative treatment of IDA via iron supplementation requires a timely screening of iron deficiency, typically done by analyzing specific blood parameters. This however of course requires drawing a blood sample which further reduces the patients' blood volume and is in many cases stated as an inconvenient procedure.
* Measured in blood zinc protoporphyrin-IX (= ZnPP) is an established parameter to detect ID.
* This study aims to evaluate a prototype device detecting ZnPP non-invasively in the intact oral mucosa of surgical patients.
* Results from the non-invasive measurement will be compared to reference measurements of ZnPP from residual blood samples (HPLC analysis) as well as to other parameters including Hb level and iron profile (MCH [= mean corpuscular hemoglobin], MCV [= mean corpuscular volume], ferritin, transferrin, transferrin saturation, soluble transferrin receptor, CRP).

DETAILED DESCRIPTION:
The non-invasive measurements will be performed using a prototype device based on fluorescence spectroscopical techniques. In brief, light (restricted wavelengths: 407 / 425nm) will be used to excite ZnPP molecules within the blood of the oral mucosa by means of an optical fibre prob. The outgoing fluorescence emission of the excited molecules will be analyzed using a spectrometer and converted to a ZnPP value [unit: µmol/mol heme] using mathematical transformations as well as spectral fitting.

This study compares the diagnostic performance of iron deficiency based on non-invasive measurements of Zinc protoporphyrin with results based on standard laboratory procedure (i.e. ZnPP measured in whole blood sample using HPLC) and blood values assessed during clinical routine, respectively.

If results of non-invasive and reference measurement techniques yield coinciding results, the non-invasive method could provide an improved mean to detect iron deficiency and thereby to improve treatment of patients suffering from iron deficiency anemia.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years

Exclusion Criteria:

* Patients who received a blood transfusion less than 8 weeks before examination
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All patients preoperatively screened for anemia in the anemia walk-in clinic of the University Hospital Frankfurt that fit the inclusion criteria will be asked to participate in the study.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2017-03-03 (Actual); Primary Completion 2018-05-01 (Actual); Study Completion 2018-05-01 (Actual)

PRIMARY OUTCOMES:
Zinc protoporphyrin blood concentration (non-invasive measurement) | Baseline
  Using the prototype device Zinc protoporphyrin blood concentration [unit: µmol/mol heme] will be measured non-invasively in the oral mucosa.
  Concentrations will be compared (Spearman's Rho, sensitivity, specificity) with Zinc protoporphyrin measurements of whole blood samples (see outcome 2 and 3).

SECONDARY OUTCOMES:
Zinc protoporphyrin blood concentration (HPLC reference measurement) | Baseline
  Using HPLC, the analytical reference method, Zinc protoporphyrin blood concentration [unit: µmol/mol heme] will be measured in whole blood samples.
Zinc protoporphyrin blood concentration (spectroscopic measurement) | Baseline
  Using fluorescence spectroscopic methods Zinc protoporphyrin blood concentration [unit: µmol/mol heme] will be measured in whole blood samples.

OTHER OUTCOMES:
Hemoglobin | Baseline
  Hemoglobin levels [unit: g/dL] will be assessed from blood samples using standardized laboratory techniques.
  Hemoglobin levels will be compared with non-invasive Zinc protoporphyrin measurements (Spearman's Rho, sensitivity, specificity).
MCH | Baseline
  MCH (= mean corpuscular hemoglobin) [unit: pg] will be assessed from blood samples using standardized laboratory techniques.
  MCH will be compared with non-invasive Zinc protoporphyrin measurements (Spearman's Rho, sensitivity, specificity).
MCV | Baseline
  MCV (= mean cell volume) [unit: fL = femtoliter] will be assessed from blood samples using standardized laboratory techniques.
  MCV will be compared with non-invasive Zinc protoporphyrin measurements (Spearman's Rho, sensitivity, specificity).
Ferritin | Baseline
  Ferritin [unit: µg/L] will be assessed from blood samples using standardized laboratory techniques.
  Ferritin levels will be compared with non-invasive Zinc protoporphyrin measurements (Spearman's Rho, sensitivity, specificity).
CRP | Baseline
  CRP (= C-reactive protein) [unit: mg/dL] will be assessed from blood samples using standardized laboratory techniques.
  CRP will be compared with non-invasive Zinc protoporphyrin measurements (Spearman's Rho, sensitivity, specificity).
Transferrin saturation | Baseline
  Transferrin saturation [unit: %] will be assessed from blood samples using standardized laboratory techniques.
  Transferrin saturation will be compared with non-invasive Zinc protoporphyrin measurements (Spearman's Rho, sensitivity, specificity).
Soluble transferrin receptor | Baseline
  Soluble Transferrin receptor [unit: mg/L] will be assessed from blood samples using standardized laboratory techniques.
  Soluble transferrin receptor will be compared with non-invasive Zinc protoporphyrin measurements (Spearman's Rho, sensitivity, specificity).

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Meybohm, Prof. Dr., Principal Investigator — Johann Wolfgang Goethe University Hospital
Locations (1):
- Johann Wolfgang Goethe University Hospital, Frankfurt am Main, Hesse, Germany

IPD SHARING:
Plan to Share IPD: Undecided